CLINICAL TRIAL: NCT04682405
Title: A Phase II Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate Uproleselan (GMI-1271) for GI Toxicity Prophylaxis During Melphalan-Conditioned Autologous Hematopoietic Cell Transplantation (Auto-HCT) for Multiple Myeloma (MM)
Brief Title: Uproleselan (GMI-1271) for GI Toxicity Prophylaxis During Melphalan-Conditioned Autologous Hematopoietic Cell Transplantation (Auto-HCT) for Multiple Myeloma (MM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: GlycoMimetics Incorporated (Industry); The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 202103086
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Results first posted 2023-12-15 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — uproleselan; Melphalan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Uproleselan + Standard of Care Melphalan (Experimental): * On the evening of Day -3, patients will receive dose #1 of uproleselan
  * On the following morning of Day -2 (12 +/- 2 hours from prior dose), patients will receive dose #2 of uproleselan
  * On the evening of Day -2 (12 +/- 2 hours from prior dose), patients will receive dose #3 of uproleselan
  * On Day -2 following completion of dose #3 of uproleselan, the patient will be administered the conditioning dose of melphalan (200mg/m^2) as per institutional practice.
  * On the following morning of Day -1 (12 +/- 2 hours from prior dose), patients will receive dose #4 of uproleselan
  * On the evening of Day -1 (12 +/- 2 hours from prior dose), patients will receive dose #5 of uproleselan
  * On the following morning of Day 0 (12 +/- 2 hours from prior dose) patients will receive dose #6 (final dose) of uproleselan
  * On Day 0, 4 hours (+/- 2 hours) after the final dose of uproleselan, the patient will be infused with the HSC product. The patient will remain inpatient until engraftment
  Interventions: Drug: Uproleselan; Drug: Melphalan
- Placebo + Standard of Care Melphalan (Placebo Comparator): * On the evening of Day -3, patients will receive dose #1 of placebo
  * On the following morning of Day -2 (12 +/- 2 hours from prior dose), patients will receive dose #2 of placebo On the evening of Day -2 (12 +/- 2 hours from prior dose), patients will receive dose #3 of placebo.
  * On Day -2 following completion of dose #3 of placebo, the patient will be administered the conditioning dose of melphalan (200mg/m^2) as per institutional practice.
  * On the following morning of Day -1 (12 +/- 2 hours from prior dose), patients will receive dose #4 of placebo.
  * On the evening of Day -1 (12 +/- 2 hours from prior dose), patients will receive dose #5 of placebo.
  * On the following morning of Day 0 (12 +/- 2 hours from prior dose) patients will receive dose #6 (final dose) of placebo.
  * On Day 0, 4 hours (+/- 2 hours) after the final dose of placebo, the patient will be infused with the HSC product. The patient will remain inpatient until engraftment
  Interventions: Drug: Placebo; Drug: Melphalan

INTERVENTIONS:
Drug: Uproleselan — Provided by study
  Other Names: GM-1271
  Arms: Uproleselan + Standard of Care Melphalan
Drug: Placebo — Provided by study
  Arms: Placebo + Standard of Care Melphalan
Drug: Melphalan — -Standard of care

SUMMARY:
The investigators hypothesize that prophylactic E-selectin inhibition via administration of uproleselan during melphalan conditioning will reduce the gastrointestinal (GI) toxicity in multiple myeloma (MM) patients undergoing auto-transplant, as assessed via diarrhea severity scoring per CTCAE v5.0, while potentially increasing chemosensitivity of malignant MM cells to high-dose melphalan.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-confirmed multiple myeloma (MM) (per IMWG criteria).
* Undergoing first auto-HCT for MM in first partial response (PR) or better
* Conditioning regimen to be single agent melphalan (200 mg/m^2)
* Adults 18 to 75 years of age, inclusive
* ECOG performance status ≤ 2
* Mobilized ≥ 5.0 x 10^6 CD34+ cells/kg (i.e. sufficient CD34+ HSCs for one auto-HCT, with at least one back-up graft in reserve)
* Adequate bone marrow and organ function prior to stem cell mobilization as defined below:

  * Leukocytes, absolute neutrophil count, and platelets within institutional standard limits for high-dose melphalan autologous stem cell transplant
  * Total bilirubin ≤ 1.5 x ULN (unless the patient has a history of Gilbert's Syndrome, in which case, total bilirubin must be ≤ 2.5 times the ULN)
  * AST(SGOT)/ALT(SGPT) ≤ 3.0 x ULN
  * Creatinine clearance ≥ 30 mL/min by Cockcroft-Gault
  * Baseline pulmonary function test (PFT) with carbon monoxide diffusion capacity in the lung (DLCO) ≥ 50% and forced expiratory volume in 1 second (FEV1) both within institutional standard limits for high-dose melphalan autologous stem cell transplant
* The effects of uproleselan (GMI-1271) on the developing human fetus are unknown. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, prior sterilization procedure, abstinence, etc.) prior to study entry, for the duration of study participation and for 12 weeks after the completion of the study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Should a man who is participating in the study become aware that he has impregnated a partner, he must inform his treating physician immediately.
* Ability to understand and willingness to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* A history of other malignancy with the exception of malignancies for which all treatment was completed at least 2 years before registration and the patient has no evidence of disease.
* Active signs or symptoms of CNS involvement by malignancy (lumbar puncture not required). Prior history of CNS involvement is acceptable, if patient has completed treatment for CNS involvement with documented treatment response.
* Prior exposure to uproleselan (GMI-1271)
* Currently receiving any other investigational agents
* A history of allergic reactions attributed to compounds of similar chemical or biologic composition to uproleselan or melphalan
* Known active infection with hepatitis A, B (e.g., HBsAg positive), or C (e.g., anti-HCV positive), or human immunodeficiency virus
* Uncontrolled acute life-threatening bacterial, viral, or fungal infection-Myocardial infarction within 6 months of uproleselan/placebo dosing, or subject has current significant cardiovascular disease, such as uncontrolled or symptomatic arrhythmias, congestive heart failure, hemodynamic instability, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification
* Any medical, psychiatric, or other condition which, in the opinion of the investigator, unfavorably alters the risk-benefit of subject participation, is likely to interfere with trial completion, assessments, or interpretation of trial results, or otherwise would make the subject an inappropriate subject for this trial.
* Pregnant and/or breastfeeding.
* Women of childbearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective contraception during the trial and for 12 weeks following the last dose of uproleselan/placebo. Women who are postmenopausal with amenorrhea for at least 1 year prior to trial entry and follicle stimulating hormone (FSH) serum levels consistent with postmenopausal status (>28U/L) will be considered NOT of childbearing potential. Highly effective contraception includes:

  * Total abstinence with a male partner.
  * Female sterilization (has had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least 6 weeks before uproleselan/placebo. In case of oophorectomy alone, the subject would be eligible only when the reproductive status of the woman has been confirmed by follow up hormone level assessment.
  * Male sterilization (at least 6 months prior to Screening). For female subjects on the trial, the vasectomized male partner should be the sole partner for that subject.
  * BOTH of the following forms of contraception consistently used together:

    * Injected, transdermal, or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%) with the exception of intrauterine devices, which are excluded due to the risk of infection and bleeding.
    * Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with or without spermicidal foam/gel/film/cream/vaginal suppository.
    * Men who are sexually active and not willing to use condoms during the trial and for 12 weeks following the last dose of uproleselan/placebo, unless they have undergone vasectomy for sterilization (at least 6 months prior to Screening), are excluded from trial participation.
* Men who are sexually active and not willing to use condoms during the trial and for 12 weeks following the last dose of uproleselan/placebo, unless they have undergone vasectomy for sterilization (at least 6 months prior to Screening), are excluded from trial participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Stockerl-Goldstein, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- Uproleselan + Standard of Care Melphalan: Patients will receive six doses of Uproleselan intravenously. The doses will begin the evening of Day -3 and continue every 12 hours through the morning of Day 0, prior to hematopoietic stem cell transplant (auto-HCT). On the evening of Day -2, patients also receive one dose of standard of care Melphalan intravenously.
- Placebo + Standard of Care Melphalan: Patients will receive six doses of placebo intravenously. The doses will begin the evening of Day -3 and continue every 12 hours through the morning of Day 0, prior to hematopoietic stem cell transplant (auto-HCT). On the evening of Day -2, patients also receive one dose of standard of care Melphalan intravenously.
Period: Overall Study
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan
Started | 26 | 25
Completed | 26 | 24
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Median (Full Range); unit: years] | 65.5 [48 to 73] | 64 [42 to 71] | 64 [42 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 11 | 20
  Male | 17 | 14 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 26 | 25 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 26 | 23 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 25 | 51

OUTCOME MEASURES:

1. Primary Outcome: Change in Diarrhea as Assessed Per CTCAE v5.0
Description: Grade 0 is defined as no diarrhea, or no change from baseline. Grade 1 is defined as an increase of <4 stools per day over baseline; mild increase in ostomy output compared to baseline. Grade 2 is defined as an increase of 4-6 stools per day over baseline; moderate increase in ostomy output compared to baseline; limiting instrumental ADL. Grade 3 is defined as an increase of >=7 stools per day over baseline; hospitalization indicated; severe increase in ostomy output compared to baseline; limited self care ADL. Grade 4 is defined as life-threatening consequences; urgent intervention indicated. Grade 5 is defined as death.
Time Frame: From day -3 to date of discharge or day 14 (whichever is sooner) (up to be 18 days)
Population: The number of participants analyzed at each time point may differ from the overall number of participants analyzed because the data was not collected. One patient in the placebo + standard of care melphalan arm was not evaluable for the outcome measure.
Measure: Mean (Standard Deviation); unit: CTCAE grade
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan
Number analyzed (Participants) | 26 | 24
CTCAE grade
  Day -3: number analyzed (Participants) | 25 | 24
  Day -3 | 0.00 (0.00) | 0.13 (0.34)
  Day -2 | 0.00 (0.00) | 0.13 (0.34)
  Day -1 | 0.31 (0.55) | 0.38 (0.58)
  Day 0 | 0.19 (0.40) | 0.21 (0.41)
  Day 1 | 0.23 (0.51) | 0.25 (0.53)
  Day 2 | 0.42 (0.58) | 0.46 (0.66)
  Day 3 | 0.65 (0.75) | 0.88 (0.85)
  Day 4 | 0.88 (0.71) | 1.08 (1.02)
  Day 5 | 1.00 (0.75) | 1.29 (0.55)
  Day 6 | 1.19 (0.85) | 1.42 (0.97)
  Day 7 | 1.42 (0.95) | 1.38 (0.77)
  Day 8 | 1.38 (0.85) | 1.63 (0.92)
  Day 9 | 1.54 (0.86) | 1.54 (0.93)
  Day 10 | 1.54 (0.86) | 1.92 (0.97)
  Day 11 | 1.46 (1.07) | 1.63 (0.92)
  Day 12 | 1.23 (0.95) | 1.17 (0.92)
  Day 13: number analyzed (Participants) | 26 | 23
  Day 13 | 1.00 (0.98) | 1.13 (0.76)
  Day 14: number analyzed (Participants) | 25 | 22
  Day 14 | 0.92 (0.76) | 0.95 (0.72)

2. Secondary Outcome: Change in Oral Mucositis as Assessed Per CTCAE v5.0
Description: Grade 0 oral mucositis is defined as no presence of mucositis. Grade 1 oral mucositis is defined as asymptomatic or mild symptoms; intervention not indicated. Grade 2 oral mucositis is defined as moderate pain or ulcer that does not interfere with oral intake; modified diet indicated. Grade 3 oral mucositis is defined as severe pain; interfering with oral intake. Grade 4 oral mucositis is defined as life-threatening consequences; urgent intervention indicated. Grade 5 oral mucositis is defined as death.
Time Frame: From day -3 to date of discharge or day 14 (whichever is sooner) (up to be 18 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CTCAE grade
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan
Number analyzed (Participants) | 26 | 24
CTCAE grade
  Day -3: number analyzed (Participants) | 25 | 24
  Day -3 | 0.00 (0.00) | 0.04 (0.20)
  Day -2 | 0.00 (0.00) | 0.04 (0.20)
  Day -1 | 0.00 (0.00) | 0.00 (0.00)
  Day 0 | 0.00 (0.00) | 0.08 (0.28)
  Day 1 | 0.00 (0.00) | 0.08 (0.28)
  Day 2 | 0.12 (0.33) | 0.08 (0.28)
  Day 3 | 0.16 (0.33) | 0.04 (0.20)
  Day 4 | 0.08 (0.27) | 0.08 (0.28)
  Day 5 | 0.12 (0.33) | 0.04 (0.20)
  Day 6 | 0.12 (0.43) | 0.17 (0.48)
  Day 7 | 0.31 (0.62) | 0.42 (0.88)
  Day 8 | 0.23 (0.51) | 0.33 (0.70)
  Day 9 | 0.38 (0.64) | 0.38 (0.71)
  Day 10 | 0.35 (0.56) | 0.33 (0.70)
  Day 11 | 0.27 (0.53) | 0.38 (0.65)
  Day 12 | 0.15 (0.46) | 0.21 (0.51)
  Day 13: number analyzed (Participants) | 26 | 23
  Day 13 | 0.15 (0.54) | 0.22 (0.52)
  Day 14: number analyzed (Participants) | 25 | 22
  Day 14 | 0.04 (0.20) | 0.23 (0.53)

3. Secondary Outcome: Change in Esophagitis as Assessed Per CTCAE v5.0
Description: Grade 0 esophagitis is defined as no presence of esophagitis. Grade 1 esophagitis is defined as asymptomatic; clinical or diagnostic observations only; intervention not indicated. Grade 2 esophagitis is defined as symptomatic; altered GI function; limiting instrumental ADL. Grade 3 esophagitis is defined as severely altered GI function; TPN indicated; elective invasive intervention indicated; limiting self care ADL. Grade 4 esophagitis is defined as life-threatening consequences; urgent operative intervention indicated. Grade 5 esophagitis is defined as death.
Time Frame: From day -3 to date of discharge or day 14 (whichever is sooner) (up to be 18 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CTCAE grade
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan
Number analyzed (Participants) | 26 | 24
CTCAE grade
  Day -3: number analyzed (Participants) | 25 | 24
  Day -3 | 0.00 (0.00) | 0.00 (0.00)
  Day -2 | 0.00 (0.00) | 0.00 (0.00)
  Day -1 | 0.00 (0.00) | 0.00 (0.00)
  Day 0 | 0.00 (0.00) | 0.00 (0.00)
  Day 1 | 0.00 (0.00) | 0.00 (0.00)
  Day 2 | 0.08 (0.27) | 0.00 (0.00)
  Day 3 | 0.04 (0.20) | 0.00 (0.00)
  Day 4 | 0.04 (0.20) | 0.04 (0.20)
  Day 5 | 0.04 (0.20) | 0.04 (0.20)
  Day 6 | 0.12 (0.43) | 0.17 (0.48)
  Day 7 | 0.23 (0.71) | 0.25 (0.68)
  Day 8 | 0.58 (1.03) | 0.25 (0.61)
  Day 9 | 0.54 (0.90) | 0.25 (0.61)
  Day 10 | 0.46 (0.86) | 0.25 (0.61)
  Day 11 | 0.38 (0.80) | 0.29 (0.62)
  Day 12 | 0.19 (0.57) | 0.21 (0.51)
  Day 13: number analyzed (Participants) | 26 | 23
  Day 13 | 0.12 (0.43) | 0.13 (0.34)
  Day 14: number analyzed (Participants) | 25 | 22
  Day 14 | 0.04 (0.20) | 0.14 (0.35)

4. Secondary Outcome: Change in Gastritis as Assessed Per CTCAE v5.0
Description: Grade 0 gastritis is defined as no presence of esophagitis. Grade 1 gastritis is defined as asymptomatic; clinical or diagnostic observations only; intervention not indicated. Grade 2 gastritis is defined as symptomatic; altered GI function; medical intervention indicated. Grade 3 gastritis is defined as severely altered eating or gastric function; TPN or hospitalization indicated. Grade 4 gastritis is defined as life-threatening consequences; urgent operative intervention indicated. Grade 5 gastritis is defined as death.
Time Frame: From day -3 to date of discharge or day 14 (whichever is sooner) (up to be 18 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CTCAE grade
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan
Number analyzed (Participants) | 26 | 24
CTCAE grade
  Day -3: number analyzed (Participants) | 25 | 24
  Day -3 | 0.00 (0.00) | 0.00 (0.00)
  Day -2 | 0.00 (0.00) | 0.00 (0.00)
  Day -1 | 0.00 (0.00) | 0.00 (0.00)
  Day 0 | 0.00 (0.00) | 0.00 (0.00)
  Day 1 | 0.04 (0.20) | 0.04 (0.20)
  Day 2 | 0.15 (0.46) | 0.13 (0.45)
  Day 3 | 0.00 (0.00) | 0.08 (0.41)
  Day 4 | 0.00 (0.00) | 0.04 (0.20)
  Day 5 | 0.00 (0.00) | 0.04 (0.20)
  Day 6 | 0.08 (0.39) | 0.08 (0.28)
  Day 7 | 0.12 (0.59) | 0.08 (0.41)
  Day 8 | 0.19 (0.63) | 0.04 (0.21)
  Day 9 | 0.23 (0.65) | 0.09 (0.29)
  Day 10 | 0.19 (0.63) | 0.13 (0.45)
  Day 11 | 0.12 (0.59) | 0.17 (0.48)
  Day 12 | 0.08 (0.39) | 0.13 (0.34)
  Day 13: number analyzed (Participants) | 26 | 23
  Day 13 | 0.04 (0.20) | 0.09 (0.29)
  Day 14: number analyzed (Participants) | 25 | 22
  Day 14 | 0.00 (0.00) | 0.05 (0.21)

5. Secondary Outcome: Change in Esophageal Pain as Assessed Per CTCAE v5.0
Description: Grade 0 esophageal pain is defined as no esophageal pain. Grade 1 esophageal pain is defined as mild pain. Grade 2 esophageal pain is defined as moderate pain; limiting instrumental ADL. Grade 3 esophageal pain is defined as severe pain; limiting self care ADL. There is no grade 4 or 5 esophageal pain defined in the CTCAE v5.0.
Time Frame: From day -3 to date of discharge or day 14 (whichever is sooner) (up to be 18 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CTCAE grade
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan
Number analyzed (Participants) | 26 | 24
CTCAE grade
  Day -3: number analyzed (Participants) | 25 | 24
  Day -3 | 0.00 (0.00) | 0.00 (0.00)
  Day -2 | 0.00 (0.00) | 0.00 (0.00)
  Day -1 | 0.00 (0.00) | 0.00 (0.00)
  Day 0 | 0.00 (0.00) | 0.04 (0.20)
  Day 1 | 0.00 (0.00) | 0.04 (0.20)
  Day 2 | 0.12 (0.33) | 0.04 (0.20)
  Day 3 | 0.04 (0.20) | 0.04 (0.20)
  Day 4 | 0.08 (0.27) | 0.13 (0.34)
  Day 5 | 0.04 (0.20) | 0.13 (0.34)
  Day 6 | 0.19 (0.49) | 0.29 (0.75)
  Day 7 | 0.35 (0.80) | 0.46 (0.88)
  Day 8 | 0.46 (0.81) | 0.33 (0.76)
  Day 9 | 0.46 (0.71) | 0.29 (0.69)
  Day 10 | 0.38 (0.64) | 0.33 (0.76)
  Day 11 | 0.31 (0.55) | 0.25 (0.61)
  Day 12 | 0.19 (0.49) | 0.17 (0.56)
  Day 13: number analyzed (Participants) | 26 | 23
  Day 13 | 0.23 (0.59) | 0.13 (0.46)
  Day 14: number analyzed (Participants) | 25 | 22
  Day 14 | 0.00 (0.00) | 0.14 (0.47)

6. Secondary Outcome: Change in Abdominal Pain as Assessed Per CTCAE v5.0
Description: Grade 0 abdominal pain is defined as no abdominal pain. Grade 1 abdominal pain is defined as mild pain. Grade 2 abdominal pain is defined as moderate pain; limiting instrumental ADL. Grade 3 abdominal pain is defined as severe pain; limiting self care ADL. There is no grade 4 or 5 abdominal pain defined in the CTCAE v5.0.
Time Frame: From day -3 to date of discharge or day 14 (whichever is sooner) (up to be 18 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CTCAE grade
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan
Number analyzed (Participants) | 26 | 24
CTCAE grade
  Day -3: number analyzed (Participants) | 25 | 24
  Day -3 | 0.00 (0.00) | 0.04 (0.20)
  Day -2 | 0.00 (0.00) | 0.00 (0.00)
  Day -1 | 0.00 (0.00) | 0.04 (0.20)
  Day 0: number analyzed (Participants) | 25 | 24
  Day 0 | 0.16 (0.37) | 0.04 (0.20)
  Day 1 | 0.19 (0.40) | 0.17 (0.38)
  Day 2 | 0.35 (0.56) | 0.25 (0.44)
  Day 3 | 0.12 (0.33) | 0.13 (0.34)
  Day 4 | 0.12 (0.33) | 0.25 (0.61)
  Day 5 | 0.08 (0.27) | 0.13 (0.34)
  Day 6 | 0.31 (0.68) | 0.21 (0.41)
  Day 7 | 0.35 (0.63) | 0.29 (0.46)
  Day 8 | 0.58 (0.70) | 0.54 (0.88)
  Day 9 | 0.54 (0.81) | 0.50 (0.98)
  Day 10 | 0.38 (0.64) | 0.46 (0.78)
  Day 11 | 0.15 (0.37) | 0.38 (0.65)
  Day 12 | 0.23 (0.43) | 0.29 (0.62)
  Day 13: number analyzed (Participants) | 26 | 23
  Day 13 | 0.12 (0.33) | 0.22 (0.42)
  Day 14: number analyzed (Participants) | 25 | 22
  Day 14 | 0.12 (0.33) | 0.05 (0.21)

7. Secondary Outcome: Change in Nausea as Assessed Per CTCAE v5.0
Description: Grade 0 nausea is defined as no nausea. Grade 1 nausea is defined as loss of appetite without alteration in eating habits. Grade 2 nausea is defined as oral intake decreased without significant weight loss, dehydration or malnutrition. Grade 3 nausea is defined as inadequate oral caloric or fluid intake; tube feeding, TPN, or hospitalization indicated. There is no grade 4 or 5 nausea defined in the CTCAE v5.0.
Time Frame: From day -3 to date of discharge or day 14 (whichever is sooner) (up to be 18 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CTCAE grade
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan
Number analyzed (Participants) | 26 | 24
CTCAE grade
  Day -3: number analyzed (Participants) | 25 | 24
  Day -3 | 0.00 (0.00) | 0.08 (0.28)
  Day -2 | 0.00 (0.00) | 0.08 (0.28)
  Day -1 | 0.12 (0.33) | 0.21 (0.51)
  Day 0 | 0.35 (0.63) | 0.42 (0.72)
  Day 1 | 0.62 (0.75) | 0.63 (0.82)
  Day 2 | 1.04 (0.82) | 1.13 (0.95)
  Day 3 | 1.00 (0.80) | 0.92 (0.88)
  Day 4 | 1.00 (0.80) | 1.17 (0.82)
  Day 5 | 0.92 (0.63) | 1.29 (0.86)
  Day 6 | 1.23 (0.82) | 1.33 (0.76)
  Day 7 | 1.35 (0.80) | 1.42 (0.88)
  Day 8 | 1.23 (0.91) | 1.21 (0.93)
  Day 9 | 1.19 (0.85) | 1.38 (1.01)
  Day 10 | 1.08 (0.84) | 1.42 (1.02)
  Day 11 | 0.65 (0.80) | 1.29 (0.95)
  Day 12 | 0.62 (0.80) | 1.00 (0.98)
  Day 13: number analyzed (Participants) | 26 | 23
  Day 13 | 0.65 (0.85) | 0.83 (0.98)
  Day 14: number analyzed (Participants) | 25 | 22
  Day 14 | 0.20 (0.41) | 0.59 (0.96)

8. Secondary Outcome: Change in Vomiting as Assessed Per CTCAE v5.0
Description: Grade 0 vomiting is defined as no vomiting. Grade 1 vomiting is defined as intervention not indicated. Grade 2 vomiting is defined as outpatient IV hydration; medical intervention indicated. Grade 3 vomiting is defined as tube feeding, TPN, or hospitalization indicated. Grade 4 vomiting is defined as life-threatening consequences. Grade 5 vomiting is defined as death.
Time Frame: From day -3 to date of discharge or day 14 (whichever is sooner) (up to be 18 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CTCAE grade
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan
Number analyzed (Participants) | 26 | 24
CTCAE grade
  Day -3: number analyzed (Participants) | 25 | 24
  Day -3 | 0.00 (0.00) | 0.00 (0.00)
  Day -2 | 0.00 (0.00) | 0.00 (0.00)
  Day -1 | 0.04 (0.20) | 0.08 (0.41)
  Day 0 | 0.12 (0.43) | 0.29 (0.62)
  Day 1 | 0.27 (0.60) | 0.29 (0.62)
  Day 2 | 0.35 (0.69) | 0.63 (0.82)
  Day 3 | 0.15 (0.46) | 0.50 (0.83)
  Day 4 | 0.15 (0.46) | 0.67 (0.92)
  Day 5 | 0.19 (0.57) | 0.54 (0.78)
  Day 6 | 0.19 (0.49) | 0.46 (0.83)
  Day 7 | 0.46 (0.86) | 0.67 (0.92)
  Day 8 | 0.62 (0.94) | 0.42 (0.78)
  Day 9 | 0.42 (0.70) | 0.42 (0.78)
  Day 10 | 0.19 (0.49) | 0.38 (0.77)
  Day 11 | 0.15 (0.54) | 0.38 (0.77)
  Day 12 | 0.08 (0.28) | 0.29 (0.62)
  Day 13: number analyzed (Participants) | 26 | 23
  Day 13 | 0.00 (0.00) | 0.13 (0.46)
  Day 14: number analyzed (Participants) | 25 | 22
  Day 14 | 0.12 (0.44) | 0.09 (0.43)

9. Secondary Outcome: Change in Enterocolitis as Assessed Per CTCAE v5.0
Description: Grade 0 enterocolitis is defined as no enterocolitis. Grade 1 enterocolitis is defined as asymptomatic; clinical or diagnostic observations only; intervention not indicated. Grade 2 enterocolitis is defined as abdominal pain; mucus or blood in stool. Grade 3 enterocolitis is defined as severe or persistent abdominal pain; fever; ileus; peritoneal signs. Grade 4 enterocolitis is defined as life-threatening consequences; urgent intervention indicated. Grade 5 enterocolitis is defined as death.
Time Frame: From day -3 to date of discharge or day 14 (whichever is sooner) (up to be 18 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CTCAE grade
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan
Number analyzed (Participants) | 26 | 24
CTCAE grade
  Day -3: number analyzed (Participants) | 25 | 24
  Day -3 | 0.00 (0.00) | 0.00 (0.00)
  Day -2 | 0.00 (0.00) | 0.00 (0.00)
  Day -1 | 0.00 (0.00) | 0.00 (0.00)
  Day 0 | 0.00 (0.00) | 0.00 (0.00)
  Day 1 | 0.08 (0.27) | 0.04 (0.20)
  Day 2 | 0.04 (0.20) | 0.08 (0.41)
  Day 3 | 0.00 (0.00) | 0.00 (0.00)
  Day 4 | 0.04 (0.20) | 0.04 (0.20)
  Day 5 | 0.00 (0.00) | 0.04 (0.20)
  Day 6 | 0.00 (0.00) | 0.08 (0.28)
  Day 7 | 0.12 (0.33) | 0.08 (0.28)
  Day 8 | 0.27 (0.67) | 0.25 (0.61)
  Day 9 | 0.27 (0.60) | 0.38 (0.61)
  Day 10 | 0.23 (0.59) | 0.38 (0.82)
  Day 11 | 0.12 (0.43) | 0.25 (0.61)
  Day 12 | 0.08 (0.39) | 0.25 (0.61)
  Day 13: number analyzed (Participants) | 26 | 23
  Day 13 | 0.04 (0.20) | 0.13 (0.34)
  Day 14: number analyzed (Participants) | 25 | 22
  Day 14 | 0.00 (0.00) | 0.05 (0.21)

10. Secondary Outcome: Change in Proctitis as Assessed Per CTCAE v5.0
Description: Grade 0 proctitis is defined as no proctitis. Grade 1 proctitis is defined as rectal discomfort, intervention not indicated. Grade 2 proctitis is defined as symptomatic (e.g., rectal discomfort, passing blood or mucus); medical intervention indicated; limiting instrumental ADL. Grade 3 proctitis is defined as severe symptoms; fecal urgency or stool incontinence; limiting self-care ADL. Grade 4 proctitis is defined as life-threatening consequences; urgent intervention indicated. Grade 5 proctitis is defined as death.
Time Frame: From day -3 to date of discharge or day 14 (whichever is sooner) (up to be 18 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CTCAE grade
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan
Number analyzed (Participants) | 26 | 24
CTCAE grade
  Day -3: number analyzed (Participants) | 25 | 24
  Day -3 | 0.00 (0.00) | 0.00 (0.00)
  Day -2 | 0.00 (0.00) | 0.00 (0.00)
  Day -1 | 0.00 (0.00) | 0.00 (0.00)
  Day 0 | 0.00 (0.00) | 0.00 (0.00)
  Day 1 | 0.00 (0.00) | 0.00 (0.00)
  Day 2 | 0.04 (0.20) | 0.00 (0.00)
  Day 3 | 0.00 (0.00) | 0.00 (0.00)
  Day 4 | 0.00 (0.00) | 0.04 (0.20)
  Day 5 | 0.00 (0.00) | 0.04 (0.20)
  Day 6 | 0.12 (0.43) | 0.04 (0.20)
  Day 7 | 0.00 (0.00) | 0.04 (0.20)
  Day 8 | 0.00 (0.00) | 0.00 (0.00)
  Day 9 | 0.08 (0.27) | 0.08 (0.41)
  Day 10 | 0.08 (0.39) | 0.08 (0.41)
  Day 11 | 0.00 (0.00) | 0.00 (0.00)
  Day 12: number analyzed (Participants) | 25 | 24
  Day 12 | 0.00 (0.00) | 0.00 (0.00)
  Day 13: number analyzed (Participants) | 26 | 23
  Day 13 | 0.00 (0.00) | 0.00 (0.00)
  Day 14: number analyzed (Participants) | 25 | 22
  Day 14 | 0.00 (0.00) | 0.00 (0.00)

11. Secondary Outcome: Change in Hemorrhoids as Assessed Per CTCAE v5.0
Description: Grade 0 hemorrhoids is defined as no hemorrhoids. Grade 1 hemorrhoids is defined as asymptomatic; clinical or diagnostic observations only; intervention not indicated. Grade 2 hemorrhoids is defined as symptomatic; banding or medical intervention indicated. Grade 3 hemorrhoids is defined as severe symptoms; invasive intervention indicated. There is no grade 4 or 5 hemorrhoids defined in the CTCAE v5.0.
Time Frame: From day -3 to date of discharge or day 14 (whichever is sooner) (up to be 18 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: CTCAE grade
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan
Number analyzed (Participants) | 26 | 24
CTCAE grade
  Day -3: number analyzed (Participants) | 25 | 24
  Day -3 | 0.00 (0.00) | 0.00 (0.00)
  Day -2 | 0.00 (0.00) | 0.00 (0.00)
  Day -1 | 0.00 (0.00) | 0.00 (0.00)
  Day 0 | 0.04 (0.20) | 0.00 (0.00)
  Day 1 | 0.04 (0.20) | 0.00 (0.00)
  Day 2 | 0.08 (0.27) | 0.00 (0.00)
  Day 3 | 0.08 (0.39) | 0.00 (0.00)
  Day 4 | 0.12 (0.43) | 0.04 (0.20)
  Day 5 | 0.12 (0.43) | 0.08 (0.28)
  Day 6 | 0.15 (0.46) | 0.08 (0.28)
  Day 7 | 0.08 (0.27) | 0.08 (0.28)
  Day 8 | 0.08 (0.27) | 0.04 (0.20)
  Day 9 | 0.15 (0.37) | 0.08 (0.28)
  Day 10 | 0.12 (0.33) | 0.08 (0.28)
  Day 11 | 0.15 (0.37) | 0.04 (0.20)
  Day 12: number analyzed (Participants) | 25 | 24
  Day 12 | 0.16 (0.37) | 0.08 (0.28)
  Day 13: number analyzed (Participants) | 26 | 22
  Day 13 | 0.04 (0.20) | 0.09 (0.29)
  Day 14: number analyzed (Participants) | 25 | 22
  Day 14 | 0.08 (0.28) | 0.09 (0.29)

12. Secondary Outcome: Time to Neutrophil Engraftment
Description: -Defined as ANC ≥0.5 x 10^9/L for 3 consecutive days or ≥1.0 x 10^9/L for 1 day
Time Frame: Through date of discharge (up to be 18 days)
Population: One subject dropped out of Placebo + Standard of Care Melphalan arm due to adverse events and was not included in the analysis for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan
Number analyzed (Participants) | 26 | 24
Days | 12.77 (0.76) | 12.50 (0.98)

13. Secondary Outcome: Change in Nutritional Status as Assessed by Total Parenteral Nutrition (TPN) Days
Time Frame: Before conditioning and at day +14 or date of discharge (whichever is sooner) (up to be 18 days)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan
Number analyzed (Participants) | 26 | 24
Days | 0.19 (0.98) | 0.00 (0.00)

14. Secondary Outcome: Duration of Hospital Length of Stay
Time Frame: From date of admission for auto-HCT to date of discharge (up to be 18 days)
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan
Number analyzed (Participants) | 26 | 24
Days | 18.42 (1.98) | 18.46 (1.84)

15. Secondary Outcome: Change in Bristol Stool Scale
Description: Change in Bristol Stool Scale as measured by incidence of Type 7 Bristol Stool Scale: liquid consistency with no solid pieces.
Time Frame: From day -3 to date of discharge or day 14 (whichever is sooner) (up to be 18 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan
Number analyzed (Participants) | 26 | 24
Participants
  Day -3, AM: number analyzed (Participants) | 23 | 24
  Day -3, AM | 0 | 1
  Day -3, PM | 0 | 1
  Day -2, AM | 0 | 2
  Day -2, PM | 0 | 1
  Day -1, AM | 1 | 0
  Day -1, PM | 0 | 1
  Day 0, AM | 1 | 3
  Day 0, PM | 0 | 1
  Day 1, AM | 5 | 4
  Day 1, PM | 1 | 3
  Day 2, AM | 3 | 5
  Day 2, PM: number analyzed (Participants) | 25 | 24
  Day 2, PM | 2 | 6
  Day 3, AM | 11 | 8
  Day 3, PM: number analyzed (Participants) | 25 | 24
  Day 3, PM | 5 | 10
  Day 4, AM | 8 | 12
  Day 4, PM | 4 | 11
  Day 5, AM | 7 | 12
  Day 5, PM | 6 | 10
  Day 6, AM | 12 | 11
  Day 6, PM | 12 | 11
  Day 7, AM | 14 | 10
  Day 7, PM | 15 | 12
  Day 8, AM | 14 | 15
  Day 8, PM | 19 | 14
  Day 9, AM | 18 | 16
  Day 9, PM | 13 | 17
  Day 10, AM | 13 | 16
  Day 10, PM | 10 | 19
  Day 11, AM: number analyzed (Participants) | 25 | 24
  Day 11, AM | 9 | 19
  Day 11, PM: number analyzed (Participants) | 25 | 24
  Day 11, PM | 8 | 11
  Day 12, AM | 11 | 9
  Day 12, PM: number analyzed (Participants) | 26 | 23
  Day 12, PM | 8 | 7
  Day 13, AM: number analyzed (Participants) | 26 | 23
  Day 13, AM | 6 | 7
  Day 13, PM: number analyzed (Participants) | 25 | 22
  Day 13, PM | 3 | 8
  Day 14, AM: number analyzed (Participants) | 24 | 22
  Day 14, AM | 3 | 7
  Day 14, PM: number analyzed (Participants) | 20 | 16
  Day 14, PM | 2 | 4

16. Secondary Outcome: Change in Nutritional Status as Assessed by Change in Standing Weight
Description: Patient standing weight in kilograms was taken at specific time points to assess any changes in nutritional status.
Time Frame: Day -3, Day 8, and date of discharge or Day 14 (whichever is sooner) (up to be 18 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan
Number analyzed (Participants) | 25 | 24
kilograms
  Day -3 | 93.26 (23.22) | 89.48 (22.37)
  Day 8: number analyzed (Participants) | 24 | 23
  Day 8 | 92.81 (22.43) | 87.24 (20.67)
  Day 14 or day of discharge, whichever is sooner | 93.34 (24.11) | 89.44 (20.58)

17. Secondary Outcome: Incidence of Infection Assessed by Rates of Bacteremia (With Organism Reported When Available)
Time Frame: Through date of discharge (upto be 18 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan
Number analyzed (Participants) | 26 | 24
Participants | 8 | 5

18. Secondary Outcome: Time to First Antibiotics
Description: Measured by the time in days to the first antibiotic dose for bacteremia.
Time Frame: Through date of discharge (up to be day 18)
Population: as for outcome 1
Measure: Median (Full Range); unit: days
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan
Number analyzed (Participants) | 23 | 23
days | 10.00 [0.00 to 13.00] | 9.00 [0.00 to 12.00]

19. Secondary Outcome: Incidence of Clostridium Difficile Infections
Time Frame: Through date of discharge (up to be 18 days)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan
Number analyzed (Participants) | 26 | 24
Participants | 3 | 1

20. Secondary Outcome: Median Daily Dose of Anti-diarrheal Medications
Description: This is defined as the number of doses of anti-diarrheal medications, such as loperamide or lomotil, that participants took daily.
Time Frame: Through date of discharge (up to be 18 days)
Population: as for outcome 1
Measure: Median (Full Range); unit: number of doses in one day
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan
Number analyzed (Participants) | 23 | 21
number of doses in one day | 2.20 [1.00 to 4.33] | 2.00 [1.00 to 5.50]

21. Secondary Outcome: Median Daily Dose of Pain Medications
Description: The median daily dose of pain medications is provided as morphine equivalents.
Time Frame: Through date of discharge (up to be 18 days)
Population: as for outcome 1
Measure: Median (Full Range); unit: mg morphine equivalents
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan
Number analyzed (Participants) | 18 | 18
mg morphine equivalents | 13.02 [2.50 to 38.75] | 15.65 [5.00 to 43.39]

22. Secondary Outcome: Median Change in Scores of Patient Reported Outcomes as Measured by the CTCAE Pro Form v1.0
Description: * Questions regarding gastrointestinal toxicities
  * Responses are scored from 1-5 with 1=no symptoms to 5=severe symptoms
Time Frame: Day -3, Day +8, date of discharge or Day +14 (whichever is sooner) (up to 18 days)
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan
Number analyzed (Participants) | 25 | 24
score on a scale
  Severity of difficulty swallowing - Day -3 | 1.00 [1.00 to 3.00] | 1.00 [1.00 to 2.00]
  Severity of difficulty swallowing - Day 8: number analyzed (Participants) | 25 | 22
  Severity of difficulty swallowing - Day 8 | 1.00 [1.00 to 5.00] | 1.00 [1.00 to 5.00]
  Severity of difficulty swallowing - date of discharge or Day 14 (whichever is sooner): number analyzed (Participants) | 23 | 22
  Severity of difficulty swallowing - date of discharge or Day 14 (whichever is sooner) | 1.00 [1.00 to 3.00] | 1.00 [1.00 to 5.00]
  Severity of mouth or throat sores - Day -3 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 3.00]
  Severity of mouth or throat sores - Day 8: number analyzed (Participants) | 25 | 22
  Severity of mouth or throat sores - Day 8 | 1.00 [1.00 to 4.00] | 1.00 [1.00 to 5.00]
  Severity of mouth or throat sores - date of discharge or Day 14 (whichever is sooner): number analyzed (Participants) | 23 | 22
  Severity of mouth or throat sores - date of discharge or Day 14 (whichever is sooner) | 1.00 [1.00 to 2.00] | 1.00 [1.00 to 5.00]
  Severity of decreased appetite - Day -3 | 1.00 [1.00 to 3.00] | 1.00 [1.00 to 3.00]
  Severity of decreased appetite - Day 8: number analyzed (Participants) | 25 | 22
  Severity of decreased appetite - Day 8 | 3.00 [2.00 to 5.00] | 4.00 [1.00 to 5.00]
  Severity of decreased appetite - date of discharge or Day 14 (whichever is sooner): number analyzed (Participants) | 23 | 22
  Severity of decreased appetite - date of discharge or Day 14 (whichever is sooner) | 3.00 [1.00 to 4.00] | 3.00 [1.00 to 5.00]
  Severity of nausea - Day -3 | 1.00 [1.00 to 2.00] | 1.00 [1.00 to 3.00]
  Severity of nausea - Day 8: number analyzed (Participants) | 25 | 22
  Severity of nausea - Day 8 | 3.00 [1.00 to 5.00] | 3.50 [1.00 to 5.00]
  Severity of nausea - date of discharge or Day 14 (whichever is sooner): number analyzed (Participants) | 22 | 22
  Severity of nausea - date of discharge or Day 14 (whichever is sooner) | 2.00 [1.00 to 4.00] | 2.50 [1.00 to 5.00]
  Severity of vomiting - Day -3 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 2.00]
  Severity of vomiting - Day 8: number analyzed (Participants) | 25 | 22
  Severity of vomiting - Day 8 | 2.00 [1.00 to 4.00] | 2.00 [1.00 to 3.00]
  Severity of vomiting - date of discharge or Day 14 (whichever is sooner): number analyzed (Participants) | 23 | 22
  Severity of vomiting - date of discharge or Day 14 (whichever is sooner) | 2.00 [1.00 to 4.00] | 2.00 [1.00 to 3.00]
  Severity of heartburn - Day -3 | 1.00 [1.00 to 3.00] | 1.00 [1.00 to 3.00]
  Severity of heartburn - Day 8: number analyzed (Participants) | 25 | 22
  Severity of heartburn - Day 8 | 1.00 [1.00 to 4.00] | 1.00 [1.00 to 4.00]
  Severity of heartburn - date of discharge or Day 14 (whichever is sooner): number analyzed (Participants) | 23 | 22
  Severity of heartburn - date of discharge or Day 14 (whichever is sooner) | 1.00 [1.00 to 3.00] | 1.50 [1.00 to 4.00]
  Severity of bloating - Day -3 | 1.00 [1.00 to 3.00] | 1.00 [1.00 to 3.00]
  Severity of bloating - Day 8: number analyzed (Participants) | 25 | 22
  Severity of bloating - Day 8 | 2.00 [1.00 to 5.00] | 2.00 [1.00 to 5.00]
  Severity of bloating - date of discharge or Day 14 (whichever is sooner): number analyzed (Participants) | 23 | 22
  Severity of bloating - date of discharge or Day 14 (whichever is sooner) | 2.00 [1.00 to 3.00] | 1.50 [1.00 to 3.00]
  Severity of abdominal pain - Day -3 | 1.00 [1.00 to 3.00] | 1.00 [1.00 to 2.00]
  Severity of abdominal pain - Day 8: number analyzed (Participants) | 25 | 22
  Severity of abdominal pain - Day 8 | 2.00 [1.00 to 4.00] | 2.50 [1.00 to 4.00]
  Severity of abdominal pain - date of discharge or Day 14 (whichever is sooner): number analyzed (Participants) | 23 | 22
  Severity of abdominal pain - date of discharge or Day 14 (whichever is sooner) | 1.00 [1.00 to 3.00] | 2.00 [1.00 to 3.00]

23. Secondary Outcome: Median Change in Scores of Quality of Life as Measured by the CTCAE Pro Form v 1.0
Description: * Questions regarding gastrointestinal, pain, and psychological symptoms interfering with daily activities
  * Responses are scored from 1-5 with 1=not at all to 5=very much
Time Frame: Day -3, Day +8, date of discharge or Day +14 (whichever is sooner) (up to 18 days)
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan
Number analyzed (Participants) | 25 | 24
score on a scale
  Mouth or throat sore interference - Day -3 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 3.00]
  Mouth or throat sore interference - Day 8: number analyzed (Participants) | 25 | 22
  Mouth or throat sore interference - Day 8 | 1.00 [1.00 to 4.00] | 1.00 [1.00 to 5.00]
  Mouth or throat sore interference - date of discharge or Day 14 (whichever is sooner): number analyzed (Participants) | 23 | 22
  Mouth or throat sore interference - date of discharge or Day 14 (whichever is sooner) | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 5.00]
  Decreased appetite interference - Day -3 | 1.00 [1.00 to 3.00] | 1.00 [1.00 to 3.00]
  Decreased appetite interference - Day 8: number analyzed (Participants) | 25 | 22
  Decreased appetite interference - Day 8 | 3.00 [1.00 to 5.00] | 3.50 [1.00 to 5.00]
  Decreased appetite interference - date of discharge or Day 14 (whichever is sooner): number analyzed (Participants) | 23 | 22
  Decreased appetite interference - date of discharge or Day 14 (whichever is sooner) | 2.00 [1.00 to 5.00] | 3.00 [1.00 to 5.00]
  Abdominal pain interference - Day -3 | 1.00 [1.00 to 3.00] | 1.00 [1.00 to 2.00]
  Abdominal pain interference - Day 8: number analyzed (Participants) | 25 | 22
  Abdominal pain interference - Day 8 | 2.00 [1.00 to 4.00] | 1.50 [1.00 to 4.00]
  Abdominal pain interference - date of discharge or Day 14 (whichever is sooner): number analyzed (Participants) | 23 | 22
  Abdominal pain interference - date of discharge or Day 14 (whichever is sooner) | 1.00 [1.00 to 4.00] | 1.00 [1.00 to 4.00]
  Bowel incontinence interference - Day -3: number analyzed (Participants) | 24 | 24
  Bowel incontinence interference - Day -3 | 1.00 [1.00 to 3.00] | 1.00 [1.00 to 2.00]
  Bowel incontinence interference - Day 8: number analyzed (Participants) | 25 | 22
  Bowel incontinence interference - Day 8 | 1.00 [1.00 to 5.00] | 1.00 [1.00 to 4.00]
  Bowel incontinence interference - date of discharge or Day 14 (whichever is sooner): number analyzed (Participants) | 23 | 22
  Bowel incontinence interference - date of discharge or Day 14 (whichever is sooner) | 2.00 [1.00 to 5.00] | 1.00 [1.00 to 5.00]

24. Secondary Outcome: Median Change in Scores of Patient Reported Outcomes as Measured by the CTCAE Pro Form v1.0
Description: * Questions regarding gastrointestinal toxicities
  * Responses are scored from 1-5 with 1=never and 5=almost constantly
Time Frame: Day -3, Day +8, date of discharge or Day +14 (whichever is sooner) (up to 18 days)
Population: as for outcome 1
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan
Number analyzed (Participants) | 25 | 24
score on a scale
  Frequency of nausea - Day -3 | 1.00 [1.00 to 3.00] | 1.00 [1.00 to 4.00]
  Frequency of nausea - Day 8: number analyzed (Participants) | 25 | 22
  Frequency of nausea - Day 8 | 4.00 [1.00 to 5.00] | 4.00 [1.00 to 5.00]
  Frequency of nausea - date of discharge or Day 14 (whichever is sooner): number analyzed (Participants) | 23 | 22
  Frequency of nausea - date of discharge or Day 14 (whichever is sooner) | 3.00 [1.00 to 4.00] | 3.00 [1.00 to 5.00]
  Frequency of vomiting - Day -3 | 1.00 [1.00 to 1.00] | 1.00 [1.00 to 2.00]
  Frequency of vomiting - Day 8: number analyzed (Participants) | 25 | 22
  Frequency of vomiting - Day 8 | 2.00 [1.00 to 4.00] | 2.50 [1.00 to 4.00]
  Frequency of vomiting - date of discharge or Day 14 (whichever is sooner): number analyzed (Participants) | 23 | 21
  Frequency of vomiting - date of discharge or Day 14 (whichever is sooner) | 2.00 [1.00 to 3.00] | 2.00 [1.00 to 4.00]
  Frequency of heartburn - Day -3 | 1.00 [1.00 to 3.00] | 1.00 [1.00 to 4.00]
  Frequency of heartburn - Day 8: number analyzed (Participants) | 25 | 22
  Frequency of heartburn - Day 8 | 1.00 [1.00 to 5.00] | 1.00 [1.00 to 4.00]
  Frequency of heartburn - date of discharge or Day 14 (whichever is sooner): number analyzed (Participants) | 23 | 22
  Frequency of heartburn - date of discharge or Day 14 (whichever is sooner) | 1.00 [1.00 to 3.00] | 1.50 [1.00 to 400]
  Frequency of bloating - Day -3 | 1.00 [1.00 to 5.00] | 1.00 [1.00 to 4.00]
  Frequency of bloating - Day 8: number analyzed (Participants) | 25 | 22
  Frequency of bloating - Day 8 | 2.00 [1.00 to 5.00] | 2.00 [1.00 to 5.00]
  Frequency of bloating - date of discharge or Day 14 (whichever is sooner): number analyzed (Participants) | 22 | 22
  Frequency of bloating - date of discharge or Day 14 (whichever is sooner) | 2.00 [1.00 to 5.00] | 2.00 [1.00 to 4.00]
  Frequency of diarrhea - Day -3 | 1.00 [1.00 to 4.00] | 1.00 [1.00 to 4.00]
  Frequency of diarrhea - Day 8: number analyzed (Participants) | 25 | 22
  Frequency of diarrhea - Day 8 | 4.00 [3.00 to 5.00] | 4.00 [2.00 to 5.00]
  Frequency of diarrhea - date of discharge or Day 14 (whichever is sooner): number analyzed (Participants) | 23 | 22
  Frequency of diarrhea - date of discharge or Day 14 (whichever is sooner) | 4.00 [1.00 to 5.00] | 4.00 [1.00 to 5.00]
  Frequency of abdominal pain - Day -3 | 1.00 [1.00 to 3.00] | 1.00 [1.00 to 3.00]
  Frequency of abdominal pain - Day 8: number analyzed (Participants) | 25 | 22
  Frequency of abdominal pain - Day 8 | 2.00 [1.00 to 5.00] | 2.50 [1.00 to 5.00]
  Frequency of abdominal pain - date of discharge or Day 14 (whichever is sooner): number analyzed (Participants) | 23 | 22
  Frequency of abdominal pain - date of discharge or Day 14 (whichever is sooner) | 2.00 [1.00 to 4.00] | 2.00 [1.00 to 4.00]
  Frequency of bowel incontinence - Day -3 | 1.00 [1.00 to 3.00] | 1.00 [1.00 to 2.00]
  Frequency of bowel incontinence - Day 8: number analyzed (Participants) | 25 | 22
  Frequency of bowel incontinence - Day 8 | 2.00 [1.00 to 4.00] | 1.00 [1.00 to 4.00]
  Frequency of bowel incontinence - date of discharge or Day 14 (whichever is sooner): number analyzed (Participants) | 23 | 22
  Frequency of bowel incontinence - date of discharge or Day 14 (whichever is sooner) | 2.00 [1.00 to 5.00] | 1.50 [1.00 to 5.00]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment through D+30 post autologous hematopoietic cell transplant (auto-HCT). The median follow-up time was 47 days (full range 1-58 days). All-cause mortality was collected from start of treatment through study completion. The median follow-up time was 242 days (full range 1-536 days).
Arm/Group | Uproleselan + Standard of Care Melphalan | Placebo + Standard of Care Melphalan
All-Cause Mortality (participants affected / at risk) | 2/26 | 3/25
Serious Adverse Events (participants affected / at risk) | 5/26 | 5/25
Other Adverse Events (participants affected / at risk) | 26/26 | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Uproleselan + Standard of Care Melphalan (N=26) | Placebo + Standard of Care Melphalan (N=25)
Nausea (Gastrointestinal disorders) | 1 | 0
Fever (General disorders) | 1 | 3
Sinusitis (Infections and infestations) | 1 | 0
Bacteremia (Infections and infestations) | 1 | 0
Lung Infection (Infections and infestations) | 1 | 0
Skin Infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Uproleselan + Standard of Care Melphalan (N=26) | Placebo + Standard of Care Melphalan (N=25)
Anemia (Blood and lymphatic system disorders) | 25 | 25
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 4
Sinus Tachycardia (Cardiac disorders) | 1 | 1
Supraventricular Tachycardia (Cardiac disorders) | 0 | 1
Ear Pain (Ear and labyrinth disorders) | 0 | 1
Adrenal Insufficiency (Endocrine disorders) | 1 | 0
Eye Disorders - other (Eye disorders) | 3 | 0 — Diplopia; estropia; right eye conjunctional hemorrhage
Blurred Vision (Eye disorders) | 1 | 0
Extraocular Muscle Paresis (Eye disorders) | 1 | 0
Periorbital Edema (Eye disorders) | 2 | 0
Photophobia (Eye disorders) | 0 | 1
Vision Decreased (Eye disorders) | 1 | 0
Gastrointestinal Disorders - other (Gastrointestinal disorders) | 0 | 1 — diverticulitis
Abdominal Pain (Gastrointestinal disorders) | 21 | 18
Bloating (Gastrointestinal disorders) | 2 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 9 | 5
Diarrhea (Gastrointestinal disorders) | 26 | 24
Dry Mouth (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 9 | 7
Esophageal Pain (Gastrointestinal disorders) | 13 | 10
Esophagitis (Gastrointestinal disorders) | 10 | 7
Flatulence (Gastrointestinal disorders) | 2 | 0
Gastric Hemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 6 | 4
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 3 | 1
Hemorrhoids (Gastrointestinal disorders) | 5 | 3
Mucositis oral (Gastrointestinal disorders) | 13 | 8
Nausea (Gastrointestinal disorders) | 25 | 24
Oral Pain (Gastrointestinal disorders) | 0 | 1
Proctitis (Gastrointestinal disorders) | 4 | 2
Toothache (Gastrointestinal disorders) | 1 | 0
Typhlitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 17 | 20
Localized Edema (General disorders) | 1 | 0 — Ear
Chills (General disorders) | 1 | 2
Edema Limbs (General disorders) | 4 | 5
Facial Pain (General disorders) | 1 | 0
Fatigue (General disorders) | 23 | 20
Fever (General disorders) | 9 | 11
Generalized Edema (General disorders) | 1 | 1
Infusion Site Extravasation (General disorders) | 2 | 0
Malaise (General disorders) | 9 | 7
Neck Edema (General disorders) | 0 | 1
Non-cardiac Chest Pain (General disorders) | 1 | 1
Pain (General disorders) | 0 | 1
Allergic Reaction (Immune system disorders) | 0 | 2
Infections and Infestations - other (Infections and infestations) | 3 | 3 — Klebsiella pneumoniae; MSSA/Staph lugdunensis; Streptococcus salivarius; Streptococcus dysgalactiae; viral dermatitis; herpes simplex virus; Klebsiella pneumoniae bacteremia
Bacteremia (Infections and infestations) | 1 | 2
Enterocolitis Infectious (Infections and infestations) | 3 | 1
Folliculitis (Infections and infestations) | 0 | 1
Lung Infection (Infections and infestations) | 1 | 0
Otitis Externa (Infections and infestations) | 1 | 0
Papulopustular Rash (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 2
Skin Infection (Infections and infestations) | 3 | 1
Thrush (Infections and infestations) | 7 | 7
Urinary Tract Infection (Infections and infestations) | 1 | 0
Bruising (Injury, poisoning and procedural complications) | 2 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 2
Activated partial thromboplastin time prolonged (Investigations) | 3 | 3
Alanine aminotransferase increased (Investigations) | 3 | 4
Alkaline phosphatase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 3
Blood bilirubin increased (Investigations) | 3 | 1
Creatinine increased (Investigations) | 2 | 3
INR increased (Investigations) | 21 | 10
Lymphocyte count decreased (Investigations) | 24 | 24
Lymphocyte count increased (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 26 | 24
Platelet count decreased (Investigations) | 26 | 23
White blood cell decreased (Investigations) | 26 | 25
Anorexia (Metabolism and nutrition disorders) | 4 | 8
Dehydration (Metabolism and nutrition disorders) | 3 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 5
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 4
Hypernatremia (Metabolism and nutrition disorders) | 2 | 6
Hyperphosphatemia (Metabolism and nutrition disorders) | 2 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 23 | 23
Hypocalcemia (Metabolism and nutrition disorders) | 26 | 22
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalemia (Metabolism and nutrition disorders) | 18 | 19
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 3
Hyponatremia (Metabolism and nutrition disorders) | 8 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 21 | 20
Musculoskeletal and Connective Tissue Disorder - other (Musculoskeletal and connective tissue disorders) | 3 | 3 — Ankle pain; bilateral shoulder pain; groin pain; hip pain; knee pain; thumb weakness
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 3
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 2 | 3
Neoplasms benign, malignant, and unspecified (incl cysts and polyps) - other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Nervous System Disorders - other (Nervous system disorders) | 1 | 2 — "tastes buds"; numbness around mouth; Restless Leg Syndrome; Taste
Dizziness (Nervous system disorders) | 6 | 6
Dysgeusia (Nervous system disorders) | 0 | 2
Encephalopathy (Nervous system disorders) | 1 | 1
Headache (Nervous system disorders) | 2 | 6
Lethargy (Nervous system disorders) | 1 | 0
Paresthesia (Nervous system disorders) | 0 | 1
Peripheral Sensory Neuropathy (Nervous system disorders) | 2 | 4
Presyncope (Nervous system disorders) | 0 | 2
Tremor (Nervous system disorders) | 0 | 2
Vasovagal Reaction (Nervous system disorders) | 0 | 1
Psychiatric Disorders - other (Psychiatric disorders) | 1 | 0 — AMS - altered mental status
Agitation (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 2 | 2
Confusion (Psychiatric disorders) | 1 | 1
Delirium (Psychiatric disorders) | 1 | 1
Hallucinations (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 2
Restlessness (Psychiatric disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 5
Hematuria (Renal and urinary disorders) | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 1
Reproductive System and Breast Disorders - other (Reproductive system and breast disorders) | 0 | 1 — Vaginal bleeding
Testicular Pain (Reproductive system and breast disorders) | 1 | 1
Respiratory, Thoracic, and Mediastinal Disorders - other (Respiratory, thoracic and mediastinal disorders) | 1 | 0 — winded
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Skin and Subcutaneous Tissue Disorders - other (Skin and subcutaneous tissue disorders) | 2 | 0 — lump; multiple scattered moles/lesions on chest
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Hot Flashes (Vascular disorders) | 0 | 3
Hypertension (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 8 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-22): https://cdn.clinicaltrials.gov/large-docs/05/NCT04682405/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/05/NCT04682405/ICF_001.pdf